CLINICAL TRIAL: NCT03088670
Title: Evaluate Efficacy and Safety of Gosogliptin as Monotherapy and in Combination With Metformin vs. Vildagliptin as Monotherapy and in Combination With Metformin in Drug-naive Type 2 Diabetic Patients.
Brief Title: Efficacy and Safety of Gosogliptin as Monotherapy and in Combination With Metformin vs. Vildagliptin as Monotherapy and in Combination With Metformin in Drug-naive Type 2 Diabetic Patients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SatRx LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SRX-1374-02
Record Dates: First submitted 2017-03-18; First posted 2017-03-23 (Actual); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — gosogliptin; Vildagliptin; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gosogliptin treatment group (Experimental): 12 weeks of monotherapy and 24 weeks of combination with Metformin
  Interventions: Drug: Gosogliptin; Drug: Metformin
- Vildagliptin treatment group (Active Comparator): 12 weeks of monotherapy and 24 weeks of combination with Metformin
  Interventions: Drug: Vildagliptin; Drug: Metformin

INTERVENTIONS:
Drug: Gosogliptin — 20 mg per day, dose titration to 30 mg per day at Week 4 as required Administration: orally
  Arms: Gosogliptin treatment group
Drug: Vildagliptin — 50 mg per day, dose titration to 100 mg per day at Week 4 as required (50 mg twice a day) Administration: orally
  Arms: Vildagliptin treatment group
Drug: Metformin — 1000 mg per day starting Week 12 (500 mg twice a day), dose titration to 2000 mg per day at Week 16 as required (1000 mg twice a day).
  Administration: orally

SUMMARY:
To demonstrate that efficacy of Gosogliptin as Monotherapy and in Combination with Metformin is non-inferior to efficacy of Vildagliptin as Monotherapy and in combination with Metformin in the effects on glycosilated hemoglobin (HbA1c) at Week 12 and Week 36 compared to baseline (Week 0).

DETAILED DESCRIPTION:
* Screening of patients at Week -2
* Training for all complying patients in Diabetes Program School at Week -1 with glucometer and patient diary distribution for SMBG
* Randomization in one of two groups in the ratio 1:1.
* The 1st stage includes 12 weeks of monotherapy with Gosogliptin or Vildagliptin.
* The 2nd stage includes 24 weeks of combination therapy with Gosogliptin and Metformin or Vildagliptin and Metformin.
* Follow-up period of 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women from 18 through 78 years
2. Confirmed clinical diagnosis of type 2 diabetes mellitus
3. Drug-naive patients or patients without hypoglycemic drug treatment at least till 12 weeks before screening
4. Patient's agreed to use adequate methods of contraception during the study
5. Body mass index 22-40 kg/m2
6. HbA1c 7.5 - 11.0%
7. FPG < 15 mmol/L
8. Signed informed consent
9. Patient's ability to follow all protocol requirements

Exclusion Criteria:

1. Pregnancy and lactation, women who plan to become pregnant during the clinical study, women of child-bearing potential (i.e. non-stylized surgically and in period of post menopause less than 2 years) without adequate methods of contraception.
2. History of type 1 diabetes mellitus and other forms
3. Severe metabolic complications of diabetes as ketoacidosis, hyperosmolar coma during 6 weeks before screening
4. Severe complication of diabetes, for instance proliferative retinopathy in active stage, autonomic neuropathy or gastroparesis
5. A known allergy, hypersensitivity or contraindications to Gosogliptin, Vildagliptin, Metformin or their components
6. Convulsive disorder; system autoimmune diseases or vascular collagenosis demanding the previous or current treatment by systemic corticosteroids, cytostatics; malignancy within the last 5 years (except for a basal-cell carcinoma);
7. Significant cardiovascular diseases within 12 months of screening including: chronic heart failure of a class III or IV (NYHA), severe arrhythmia demanding treatment with antiarrhythmics, unstable angina, myocardial infarction, heart and coronary vessels surgery, heart valves diseases, transitory ischaemic attack or stroke, uncontrolled arterial hypertension with systolic Blood Pressure > 180 mm Hg and diastolic Blood Pressure > 110 mm Hg, pulmonary embolism or deep venous thrombosis
8. A nephrotic syndrome, a chronic renal failure, serum creatinine > 1.5 mg/dL (132 µmol/L) in men and > 1.4 mg/dL (123 µmol/L) in women or GFR <60 ml/min/1.73m2
9. HBV, HCV or a liver cirrhosis; AST or ALT > 3 ULN; total bilirubin > 2 ULN
10. HIV; severe infection that can affect glycemia within 30 days of screening
11. Anemia (Hb ≤10.5 g/dL in women or ≤11.5 g/dL in men); loss of > 1 unit of blood ( 500 mL) or blood transfusion within 12 weeks of screening
12. Drugs or alcohol abuse
13. Administration of any study drug within 30 days of screening
14. Inability to read or write; unwillingness to understand and follow the protocol procedures

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2013-04-23 (Actual); Primary Completion 2014-03-30 (Actual); Study Completion 2014-10-03 (Actual)

PRIMARY OUTCOMES:
Mean change of HbA1c | at Weeks 12 and 36 from baseline
  Gosogliptin treatment group vs. Vildagliptin treatment group

SECONDARY OUTCOMES:
HbA1c level of ≤7% | at Weeks 12 and 36 from baseline
  Percent of patients who reach the target HbA1c
Hypoglycemic episodes | up to 36 week
  Incidence of hypoglycemic episodes during the monotherapy and in combination with Metformin
Fasting plasma glucose | at Weeks 12 and 36
  Change of fasting plasma glucose from baseline
Change of Body Mass | at Weeks 12 and 36
  Change of Body Mass from baseline
Adverse event | up to 40 week
  AE rate

CONTACTS AND LOCATIONS:
Locations (27):
- Russia (27):
  - Non-state healthcare Organization "Road Clinical Hospital at the station Chelyabinsk Open Joint Stock Company" Russian Railways, Chelyabinsk
  - State Budget Healthcare Institution of Moscow "Endocrinology Dispensary", Moscow
  - SEI HPE "First Moscow State Medical University n.a. I.M. Sechenov of Ministry of Health and Social Development of the Russian Federation", Chair of faculty therapy #2 based at SHI of Moscow "City clinical hospital #61", Moscow
  - State Budget Educational Institution higher professional education "1st Moscow State Medical University n.a. I.M. Sechenov of the Ministry of Healthcare of Russian Federation", Moscow
  - Federal State Institution "Clinical Hospital № 1" of the Office of the President of the Russian Federation, Moscow
  - State Budget Healthcare Institution of Moscow city "City Clinical Hospital # 71 by the Department of Healthcare in Moscow", Moscow
  - State Budget Educational Institution of higher professional education "1st Moscow State Medical University n.a. I.M. Sechenov of the Ministry of Healthcare of Russian Federation" based on Endocrinology department of Hospital № 67 n.a L A Vorohobova, Moscow
  - SEI APE "Russian Medical Academy of Postgraduate Education of Roszdrav", Chair of endocrinology and diabetology with course of endocrine surgery based at FSI "Central Clinical hospital of civil aviation", Moscow
  - State budgetary institution "Nizhny Novgorod Regional Clinical Hospital n.a Semashko, Nizhny Novgorod
  - State Health Care Institution "Perm Regional Hospital for War Veterans", Perm
  - State Educational Institution of Higher Professional Education "Perm State Medical Academy n.a. academician EA Wagner's "Ministry of Health of the Russian Federation on the basis of Department of Endocrinology Regional Clinical Hospital, Perm
  - SHI "Republic Hospital n.a. V.A. Baranov", Petrozavodsk
  - State budgetary institution of Ryazan region "City Clinical Hospital № 11", Ryazan
  - St. Petersburg State healthcare institution "City Outpatient Clinic #37", Saint Petersburg
  - FSHI "Clinical Hospital #122 n.a. L.G. Sokolov of FMBA of Russia", Internal medicine department, Saint Petersburg
  - State Health Care Institution Leningrad Regional Hospital, Saint Petersburg
  - Autonomous Noncommercial Organization "Medical Centre "XXI сentury", Saint Petersburg
  - St. Petersburg State healthcare institution "City Hospital of Saint Martyr Elizaveta", Saint Petersburg
  - FSMEI HPE "Military Medical Academy n.a. S.M. Kirov" of the Ministry of Defence of the Russian Federation, 1st Internal medicine Chair of advanced training, Saint Petersburg
  - "Diabetes Center "LLC, Samara
  - State Budget Educational Institution higher professional education "Saratov State Medical University n.a. V.I. Razumovsky" of the Ministry of Healthcare of Russian Federation based on Clinical Hospital n.a S.R. Mirotvortsev, Saratov
  - Municipal health care institution "City polyclinic №20, Saratov
  - SBEI HPE "Smolensk State Medical Academy" of the Ministry of Health and Social Development of the Russian Federation, Center of clinical research of diagnostic and medicinal products, Chair of clinical pharmacology, Smolensk
  - State budget educational institution of higher education "Smolensk State Medical Academy," of Ministry of Health and Social Development of the Russian Federation on the basis of sanatorium SSMA, Smolensk
  - State autonomous healthcare institution of Yaroslavl Region "Сlinical hospital for emergency medical care n. a. N.V. Solovyov", Yaroslavl
  - Municipal clinical health institution Health Service Novo-Yaroslavl Oil Refinery, Yaroslavl
  - SHI of Yaroslavl region "Regional Clinical Hospital", Endocrinology department, Yaroslavl

IPD SHARING:
Plan to Share IPD: No